CLINICAL TRIAL: NCT00680524
Title: Telephone Based Care for OIF/OEF Veterans With PTSD
Brief Title: Telephone-based Care for OEF/OIF Veterans With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SHP 08-184
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Results first posted 2014-09-26 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-06

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: telephone-based intervention for PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phone Based Outreach Intervention Group (Experimental): Open pilot trial
  Interventions: Other: Phone-based outreach

INTERVENTIONS:
Other: Phone-based outreach — Nurse care managers will use a phone call outreach intervention with structured templated notes to help deliver evidence-based care for PTSD

SUMMARY:
Objective: OEF/OIF (Operation Enduring Freedom and Operation Iraqi Freedom) veterans are presenting with high rates of PTSD. Translating Initiatives for Depression into Effective Solutions (TIDES) is a model of phone-based care being implemented nationally as a model to address those patients suffering from depression, PTSD, or alcohol use disorders. However, evidence-based treatments do not yet exist for phone-based management of OEF/OIF veterans who suffer from PTSD.

Research Plan:

This is an open trial to assess feasibility of augmenting standard treatment of PTSD with TIDES based telephone-based nurse care management.

DETAILED DESCRIPTION:
Background:

Veterans from Operation Enduring Freedom and Operation Iraqi Freedom (OEF/OIF) present with high rates of post-traumatic stress disorder (PTSD) and depressive disorders, but may experience barriers to specialty mental health (MH) care. Recent research suggests the majority of OEF/OIF veterans referred to MH for PTSD or depression fail to attend the recommended number of appointments within the first year. The TIDES (Translating Initiatives for Depression into Effective Solutions) model of collaborative care management for depression is an evidence-based option for VA primary care settings. However, patients in TIDES care management often have co-morbid PTSD, and the current model does not include PTSD-specific tools.

Objectives:

The primary objectives of the project were to assess feasibility and acceptability of (1) adapting TIDES tools and protocols to include PTSD and depression in the management of OEF/OIF patients, and (2) implementing the adapted model to augment treatment as usual in the VA Seattle-Puget Sound Deployment Health Clinic (DHC).

Methods:

We conducted a pilot implementation of the TIDES/PTSD model in a single site that provides integrated care specifically for OEF/OIF veterans. TIDES CPRS (Computerized Patient Record System) templates were adapted to include assessment and monitoring for PTSD. Phone-based care management protocols were expanded to include PTSD in three clinical domains: (1) medication management, (2) psychosocial support, and (3) patient self-management support, including the optional workbook "Strategies for Managing Stress After the War: Veterans Workbook." The templates were written in VA Class 1 Software, and clinical data were coded as Health Factors, allowing for automatic collection into the VISN 20 Data Warehouse. TIDES Care Managers were trained to use these templates, protocols, and workbook. Clinical staff received an orientation to the model of care. We enrolled 20 patients, newly initiating care at the DHC, who had a clinical diagnosis of PTSD and score of 50 or greater on the PTSD Check List-Military version (PCL-M). Co-morbid depression, if present, was defined by clinical diagnosis and a score of 10 or greater on the nine-item Patient Health Questionnaire (PHQ-9). Patients were followed by a Care Manager for up to six months. Formative evaluation included utilization data, clinical data, and qualitative data from semi-structured interviews of clinical staff and patients on their experiences with the model.

Status:

Final report.

ELIGIBILITY:
Inclusion Criteria:

* PTSD
* Operation Enduring Freedom and Operation Iraqi Freedom veteran

Exclusion Criteria:

* no phone
* severe brain injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradford L. Felker, MD BA, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Open pilot trial
  Phone-based outreach: Nurse care managers will use a phone call outreach intervention with structured templated notes to help deliver evidence-based care for PTSD
Period: Overall Study
Arm/Group | Arm 1
Started | 20
Completed | 17
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Acceptability to Providers and Patients
Description: Patients and providers rated the components of the intervention on a 5 point scale where 1 = poor and 5 = excellent and average ratings for each group is reported below
Time Frame: Six months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1
Number analyzed (Participants) | 20
units on a scale
  Rating of Medication support | 4.7 (.5)
  Rating of Health Education | 3.8 (1.3)
  Rating of pt self management activation | 3.8 (.5)

ADVERSE EVENTS:
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes